CLINICAL TRIAL: NCT02355418
Title: A Prospective Observational Study Examining the Role of Myocardial Fibrosis in Outcome Following Mitral Valve Repair in Degenerative Mitral Regurgitation.
Brief Title: The Role of Myocardial Fibrosis in Degenerative Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Boyang Liu, Cardiology Research Fellow, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: Not yet available
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Mitral Valve Regurgitation; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken from all patients as part of their routine care, including measurements for full blood count, urea and electrolytes, liver function test, and markers of cardiac fibrosis.
  In patients who chooses to undergo surgical repair of mitral regurgitation, myocardial biopsies will be taken to look for the degree of diffuse myocardial fibrosis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients for early surgery: A prospective, cross sectional comparison of asymptomatic patients before and after mitral valve repair surgery for chronic severe primary degenerative mitral regurgitation.Once established, it is our intention to restudy subjects in 5 years to provide information on late outcome following surgery.
  Interventions: Procedure: Mitral valve repair
- Patients against early surgery: In order to establish the natural history of diffuse fibrosis in mitral regurgitation, an additional cohort of patients with asymptomatic mitral regurgitation who do not wish to consider early repair will be followed.

INTERVENTIONS:
Procedure: Mitral valve repair — Standard mitral valve repair surgery
  Groups: Patients for early surgery

SUMMARY:
This study investigates the hypothesis that diffuse interstitial cardiac fibrosis develops in response to chronic volume overload from severe degenerative mitral regurgitation. The investigators will investigate the functional (exercise) and symptomatic (PROMS) outcomes of patients with severe but asymptomatic mitral regurgitation who have the option of choosing surgical repair or watchful waiting.

DETAILED DESCRIPTION:
The optimal management of chronic severe primary degenerative mitral regurgitation (MR) is to repair the valve, but timing of surgery remains controversial. Current guidelines suggest 'watchful waiting' until the onset of symptoms or left ventricular dysfunction but have been criticized for promoting 'rescue surgery'. Better predictors are required to optimize timing of surgery and patient outcomes.

Chronic volume overload is a stimulus for adverse adaptive left ventricular (LV) remodeling. Subclinical reduction in LV strain before mitral repair predicts a fall in LV ejection fraction following surgery and is thought to reflect myocardial fibrosis. The investigators' pilot cardiac magnetic resonance (CMR) data support this hypothesis. The aims of this study are:

1. identify whether diffuse interstitial myocardial fibrosis impacts upon post-operative complications, symptomatic improvement and ventricular recovery following surgery,
2. to show that diffuse fibrosis (assessed by T1 mapping CMR) is validated by histological assessment on myocardial biopsy,
3. identify independent pre-operative imaging / biomarker / exercise predictors of post-operative clinical outcomes

The investigators will investigate and follow up patients with severe degenerative mitral regurgitation, who do meet a class 1 indication for mitral valve surgery using present AHA guidelines. Patients have the option of choosing either close monitoring or early surgical repair of their mitral valve (class 2a indication). The relationship between patient symptoms, CMR findings, blood and histological measures of fibrosis will be studied and correlated with patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

(1) All patients with asymptomatic chronic, severe primary degenerative MR known to the Queen Elizabeth Hospital Birmingham (of note, the aetiology and severity of MR will be based on the echocardiography findings , interpreted according to the European Association of Echocardiography recommendations).

Exclusion Criteria:

1. symptoms due to severe MR;
2. LV endsystolic diameter >45mm at baseline;
3. LV ejection fraction <60%;
4. history of myocardial infarction, previous coronary artery bypass graft, or valve surgery;
5. inherited or acquired cardiomyopathy;
6. congenital heart disease; including common atrio-ventricular canal defects;
7. more than mild coexisting aortic valve stenosis or regurgitation
8. primary mitral regurgitation not due to degenerative disease, including rheumatic disease and infective endocarditis;
9. uncontrolled atrial fibrillation (resting HR>100/min average on 24 hour Holter );
10. unable to undergo CMR;
11. unable to walk on treadmill or use supine bicycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with asymptomatic chronic, severe primary degenerative mitral regurgitation (MR) under clinical follow-up or on the surgical waiting list at Queen Elizabeth Hospital Birmingham (QEHB). Aetiology and severity of MR will be based on the findings of echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Detection of diffuse interstitial fibrosis in patients with chronic severe degenerative mitral regurgitation and evaluation of its functional consequences. | 3 years
  Using T1-mapping CMR and myocardial biopsy, the investigators can confirm the development of diffuse interstitial fibrosis in patients with chronic severe degenerative mitral regurgitation. Using a range of clinical markers, the investigators will study the development of diffuse interstitial fibrosis and its relationship to left ventricular recovery following surgery, length of in-hospital stay, and patients' functional (exercise) and symptomatic (PROMS) status.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Steeds, Principal Investigator — University Hospital Birmingham
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Liu B, Neil DAH, Bhabra M, Patel R, Barker TA, Nikolaidis N, Billing JS, Hayer M, Baig S, Price AM, Vijapurapu R, Treibel TA, Edwards NC, Steeds RP. Reverse Myocardial Remodeling Following Valve Repair in Patients With Chronic Severe Primary Degenerative Mitral Regurgitation. JACC Cardiovasc Imaging. 2022 Feb;15(2):224-236. doi: 10.1016/j.jcmg.2021.07.007. Epub 2021 Aug 18. PMID 34419393
- [Derived] Liu B, Neil DAH, Premchand M, Bhabra M, Patel R, Barker T, Nikolaidis N, Billing JS, Treibel TA, Moon JC, Gonzalez A, Hodson J, Edwards NC, Steeds RP. Myocardial fibrosis in asymptomatic and symptomatic chronic severe primary mitral regurgitation and relationship to tissue characterisation and left ventricular function on cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2020 Dec 14;22(1):86. doi: 10.1186/s12968-020-00674-4. PMID 33308240
- [Derived] Liu B, Edwards NC, Neal DAH, Weston C, Nash G, Nikolaidis N, Barker T, Patel R, Bhabra M, Steeds RP. A prospective study examining the role of myocardial Fibrosis in outcome following mitral valve repair IN DEgenerative mitral Regurgitation: rationale and design of the mitral FINDER study. BMC Cardiovasc Disord. 2017 Nov 22;17(1):282. doi: 10.1186/s12872-017-0715-y. PMID 29166877